CLINICAL TRIAL: NCT04270708
Title: Intranasal Dexmedetomidine vs Oral Triclofos Sodium Sedation for Children With Autism Undergoing Electroencephalograms - A Randomized Controlled Trial.
Brief Title: Intranasal Dexmedetomidine vs Oral Triclofos Sodium for EEG in Children With Autism
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rabin Medical Center (Other)
Responsible Party: Principal Investigator, Eytan Kaplan, Director of Pediatric Sedation Services, Schneider Children's Medical Center of Israel, Rabin Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 0090-20-RMC
Record Dates: First submitted 2020-02-13; First posted 2020-02-17 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Autistic Disorder
Keywords: Sedation
MeSH Terms: conditions — Autistic Disorder | interventions — Dexmedetomidine; triclofos

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dexmedetomidine (Experimental): Intranasal Dexmedetomidine 3mcg/kg
  Interventions: Drug: Dexmedetomidine
- Triclofos (Active Comparator): Oral Triclofos Sodium 50mg/kg
  Interventions: Drug: Triclofos 100 MG/ML

INTERVENTIONS:
Drug: Dexmedetomidine — Patients with Autism will be treated with intranasal Dexmedetomidine as a sedative for EEG
  Arms: Dexmedetomidine
Drug: Triclofos 100 MG/ML — Patients with Autism will be treated with oral Triclofos as a sedative for EEG
  Arms: Triclofos

SUMMARY:
Children with Autistic Spectrum Disorder (ASD) often undergo an Electroencephalography (EEG) as part of routine work up. These children present a challenge to successful EEG execution, due to a lack of co-operation, and thus, are often in need of sedation. Historically we have used orally administered, Triclofos Sodium (TFS) - pharmacologically and physiologically similar to chloral hydrate, for sedation in this age group. However success using this drug is limited to approximately 75% in those aged 5 years and above, and possibly lower in this age group when associated with a diagnosis of ASD. The medication is often poorly tolerated by the oral route, and involves patient agitation, spiting (with incomplete drug ingestion), and immediate vomiting upon administration. Recently we have introduced Intra-nasal Dexmedetomidine (IN DEX), with an initial impression of much improved drug acceptance and possibly improved efficacy over TFS.

We designed this pilot study, with the aim of comparing efficacy, tolerance of drug administration and adverse events between TFS and IN DEX, with the goal of generating initial results as well as feasibility of recruitment for a larger trial.

DETAILED DESCRIPTION:
Study participants will be allocated, amongst patients invited for routine EEG monitoring in the hospitals EEG facility. All patients will be fasted on arrival, with a recommendation to awaken early on the day of the planned examination.

Patients aged 4yrs and above, with a diagnosis of ASD will be allocated and investigated for fulfillment of inclusion and exclusion criteria for study participation. The legal guardians of patients meeting study criteria will be approached for study participation consent. Patients declining consent will be treated with TFS as per current protocol. Patients for whom consent is attained will comprise the study group.

Study group patients will be randomized for treatment and stratified according to age groups: 4-7, 8-12, 12-18. Treatment will consist of 2 alternative pathways:

Oral Trichlofos Sodium (TFS) Pathway:

1. Initial Drug dose: Patients will be treated orally with 50mg/kg of TFS to maximum of 2000gr.
2. Failure to achieve sedate state 45 minutes after drug administration will enable an additional oral dose of 25mg/kg.
3. Patients failing to fall asleep following second drug dose will be regarded as treatment failure.
4. Rescue therapy according to physician's choice can be instituted (Dexmed or Neuleptil).

Intranasal Dexmedetomidine (IN DEX) Pathway:

1. Initial drug dose: Patients will be treated with IN 3mcg/kg of Dexmedetomidine to max dose of 150mcg. The drug will be delivered through MAD nasal atomizer.
2. Failure to achieve sedate state 45 minutes after drug administration will enable an additional dose of IN 1.5mcg/kg by MAD device.
3. Paitients failing to fall asleep following second drug dose will be regarded as treatment failure.
4. Rescue therapy according to physician's choice can be instituted (Neuleptil not recommended due to drug interactions).

All sedated children will be connected to monitoring including ECG chest leads in addition to oxygen pulse saturation monitoring.

Primary outcome assessment: Sedation depth by UMSS will be assessed by the EEG technician, who will be blinded to the drug used for sedation.

Secondary outcome assessment:

1. Satisfaction from sedation depth for completing exam by blinded technician on VAS score.
2. EEG motion artifact by interpreting neurologist, blinded to study drug on VAS score.
3. All other secondary outcomes from drug administration to discharge, including adverse events and needed interventions, will be documented by the nurse who is not blinded to administered drug.
4. ECG monitoring for determination of HR or arrhythmia
5. Assessing incidence of bradycardia, hypotension and their severity:

   a. HR and BP age related normal value chart to be used as reference. b. Bradycardia and Hypotension determined in relation to lower normal value for age: i. Mild<10% decrease from normal value ii. Moderate 10-20% decrease from normal value iii. Severe >20% or signs of hemodynamic compromise

   Ethics: This study is a comparison of two medications currently under routine use for performing sedated EEG's in our medical center. The study will be authorized by the Rabin Campus Helsinki Committee. Informed consent will be requested from the accompanying legal guardian.

   Statistics: Based on our experience, we assume a 70% success rate for sedation using TFS and a 90% success rate for IN DEX. Using an alpha of 0.05 and 80% power, two groups of 62 patients would be needed, to demonstrate statistical significance.

   This trial is planned as a pilot study aimed at assessing drug effects and recruitment rate, over a limited time period of up to 2 year, or up to 200 patiens (100 TFS + 100 IN DEX).

   Randomization and age stratification: Patient allocation will be determined according to an age stratified randomization table. Patients will be stratified by 3 age groups: 4-7, 8-12, 12-18.

   Funding: No funding has been allocated for this study. Study will be conducted using routine medications in current practice without additional cost.

ELIGIBILITY:
Inclusion Criteria:

1. Children aged 4-18 yrs referred for an EEG under sedation..
2. A Neurologist derived diagnosis of Autistic Spectrum Disorder (ASD).
3. ASA 1 or 2

Exclusion Criteria:

1. Allergy to study drug
2. Congenital heart disease, bradycardia < 60 or know arrhythmia/AV block.
3. Vasoactive drugs or treatment for arterial HTN.
4. Known Renal dysfunction Creatinine Clearance < 30% or known Liver dysfunction (Elevated LFT's).
5. Concurrent Treatment with drugs know to interact with Dexmedetomidine:

   1. Atipical Antipsychotics / Phenothiazines
   2. Tricyclic anti-depressents
   3. Lacosamide treatment - Antiepileptic.
   4. PDE V inhibitors (Viagra)
   5. Beta-blockers
   6. Phenothiazines
   7. First generation Anti-histamines
6. Significant rhinorrhea.

Ages: 3 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 200 (Estimated)
Dates: Start 2020-03-01 (Estimated); Primary Completion 2022-03-01 (Estimated); Study Completion 2022-08-01 (Estimated)

PRIMARY OUTCOMES:
Maximal Sedation Depth | Within 90 minutes
  Maximal Sedation Depth by the University of Michigan Sedation Scale (UMSS)
Technician satisfaction from sedation | Within 90 minutes
  Technician Ability to complete exam in satisfactory fashion - VAS score

SECONDARY OUTCOMES:
Neurologist satisfaction from EEG motion artifact | Within 7 days
  Neurologist satisfaction from EEG motion artifact - VAS score
Compliance with IN vs Oral Delivery | Immediate upon administration
  Compliance with IN vs Oral Delivery - Successful drug administration Y/N?
Resistance to drug administration (1-10 scale) | Immediate upon administration
  Resistance to drug administration (1-10 scale): Crying / spitting or Complete or Partial Rejection for TFS/IN DEX
Achieving sedation following single dose | Within 45 minutes
  Achieving sedation following single dose of Dexmed vs TFS
Achieving sedation following rescue dose | within 90 minutes
  Achieving sedation following additional rescue dose of Dexmed vs TFS
Sedation onset, duration and recovery periods | Within 4 hours.
  Sedation onset, duration and recovery periods
Adverse Events | Within 4 hours.
  Sedation associated adverse events

REFERENCES:
- [Result] Baio J, Wiggins L, Christensen DL, Maenner MJ, Daniels J, Warren Z, Kurzius-Spencer M, Zahorodny W, Robinson Rosenberg C, White T, Durkin MS, Imm P, Nikolaou L, Yeargin-Allsopp M, Lee LC, Harrington R, Lopez M, Fitzgerald RT, Hewitt A, Pettygrove S, Constantino JN, Vehorn A, Shenouda J, Hall-Lande J, Van Naarden Braun K, Dowling NF. Prevalence of Autism Spectrum Disorder Among Children Aged 8 Years - Autism and Developmental Disabilities Monitoring Network, 11 Sites, United States, 2014. MMWR Surveill Summ. 2018 Apr 27;67(6):1-23. doi: 10.15585/mmwr.ss6706a1. PMID 29701730
- [Result] Keller R, Basta R, Salerno L, Elia M. Autism, epilepsy, and synaptopathies: a not rare association. Neurol Sci. 2017 Aug;38(8):1353-1361. doi: 10.1007/s10072-017-2974-x. Epub 2017 Apr 28. PMID 28455770
- [Result] Thoresen M, Henriksen O, Wannag E, Laegreid L. Does a sedative dose of chloral hydrate modify the EEG of children with epilepsy? Electroencephalogr Clin Neurophysiol. 1997 Feb;102(2):152-7. doi: 10.1016/s0921-884x(96)96509-1. PMID 9060867
- [Result] Nordt SP, Rangan C, Hardmaslani M, Clark RF, Wendler C, Valente M. Pediatric chloral hydrate poisonings and death following outpatient procedural sedation. J Med Toxicol. 2014 Jun;10(2):219-22. doi: 10.1007/s13181-013-0358-z. PMID 24532346
- [Result] Sing K, Erickson T, Amitai Y, Hryhorczuk D. Chloral hydrate toxicity from oral and intravenous administration. J Toxicol Clin Toxicol. 1996;34(1):101-6. doi: 10.3109/15563659609020242. PMID 8632499
- [Result] Hirsch IA, Zauder HL. Chloral hydrate: a potential cause of arrhythmias. Anesth Analg. 1986 Jun;65(6):691-2. No abstract available. PMID 3706808
- [Result] Grissinger M. Chloral Hydrate: Is It Still Being Used? Are There Safer Alternatives? P T. 2019 Aug;44(8):444-459. PMID 31447530
- [Result] Kaplan E, Daka A, Weissbach A, Kraus D, Kadmon G, Milkh R, Nahum E. Triclofos Sodium for Pediatric Sedation in Non-Painful Neurodiagnostic Studies. Paediatr Drugs. 2019 Oct;21(5):371-378. doi: 10.1007/s40272-019-00346-6. PMID 31292919
- [Result] Mason KP, Lubisch N, Robinson F, Roskos R, Epstein MA. Intramuscular dexmedetomidine: an effective route of sedation preserves background activity for pediatric electroencephalograms. J Pediatr. 2012 Nov;161(5):927-32. doi: 10.1016/j.jpeds.2012.05.011. Epub 2012 Jun 15. PMID 22704249
- [Result] Liu H, Sun M, Zhang J, Tian Q, Yu Q, Liu Y, Yang F, Li S, Tu S. Determination of the 90% effective dose of intranasal dexmedetomidine for sedation during electroencephalography in children. Acta Anaesthesiol Scand. 2019 Aug;63(7):847-852. doi: 10.1111/aas.13372. Epub 2019 Apr 14. PMID 30982953
- [Result] Baier NM, Mendez SS, Kimm D, Velazquez AE, Schroeder AR. Intranasal dexmedetomidine: an effective sedative agent for electroencephalogram and auditory brain response testing. Paediatr Anaesth. 2016 Mar;26(3):280-5. doi: 10.1111/pan.12851. PMID 26814037
- [Result] Gumus H, Bayram AK, Poyrazoglu HG, Canpolat DG, Per H, Canpolat M, Yildiz K, Kumandas S. Comparison of Effects of Different Dexmedetomidine and Chloral Hydrate Doses Used in Sedation on Electroencephalography in Pediatric Patients. J Child Neurol. 2015 Jul;30(8):983-8. doi: 10.1177/0883073814549582. Epub 2014 Sep 22. PMID 25246305
- [Result] Fernandes ML, Oliveira WM, Santos Mdo C, Gomez RS. Sedation for electroencephalography with dexmedetomidine or chloral hydrate: a comparative study on the qualitative and quantitative electroencephalogram pattern. J Neurosurg Anesthesiol. 2015 Jan;27(1):21-5. doi: 10.1097/ANA.0000000000000077. PMID 24823763
- [Result] Kogan A, Katz J, Efrat R, Eidelman LA. Premedication with midazolam in young children: a comparison of four routes of administration. Paediatr Anaesth. 2002 Oct;12(8):685-9. doi: 10.1046/j.1460-9592.2002.00918.x. PMID 12472704
- [Result] Poonai N, Spohn J, Vandermeer B, Ali S, Bhatt M, Hendrikx S, Trottier ED, Sabhaney V, Shah A, Joubert G, Hartling L. Intranasal Dexmedetomidine for Procedural Distress in Children: A Systematic Review. Pediatrics. 2020 Jan;145(1):e20191623. doi: 10.1542/peds.2019-1623. PMID 31862730
- [Result] Li BL, Zhang N, Huang JX, Qiu QQ, Tian H, Ni J, Song XR, Yuen VM, Irwin MG. A comparison of intranasal dexmedetomidine for sedation in children administered either by atomiser or by drops. Anaesthesia. 2016 May;71(5):522-8. doi: 10.1111/anae.13407. Epub 2016 Mar 3. PMID 26936022
- [Result] Xie Z, Shen W, Lin J, Xiao L, Liao M, Gan X. Sedation effects of intranasal dexmedetomidine delivered as sprays versus drops on pediatric response to venous cannulation. Am J Emerg Med. 2017 Aug;35(8):1126-1130. doi: 10.1016/j.ajem.2017.03.021. Epub 2017 Mar 18. PMID 28347608
- [Result] Iirola T, Vilo S, Manner T, Aantaa R, Lahtinen M, Scheinin M, Olkkola KT. Bioavailability of dexmedetomidine after intranasal administration. Eur J Clin Pharmacol. 2011 Aug;67(8):825-31. doi: 10.1007/s00228-011-1002-y. Epub 2011 Feb 12. PMID 21318594